CLINICAL TRIAL: NCT04299269
Title: "Info-AF" Information Preferences in Patients With Atrial Fibrillation/Flutter and the Association With Clinical Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Nikola Schütz, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1617/2019
Record Dates: First submitted 2020-02-28; First posted 2020-03-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire including questions about Quality of life, symptoms and general informations

SUMMARY:
The aim of this project is to identify a variable that discerns patients who are interested in their disease (atrial fibrillation/atrial flutter) from patients who show no interest and furthermore test this theory in a questionnaire survey.

This should help distinguish between patients who are interested in shared decision making and patients who are not (further projects planned).

ELIGIBILITY:
Inclusion Criteria:

* Current atrial fibrillation/flutter
* >18 years of age
* sufficient knowledge of the german language to fill out the questionnaire

Exclusion Criteria:

* < 18 years of age
* insufficient knowledge of the german language to fill out the questionnaire
* Hemodynamic instability

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Preferences for autonomy measured with questionnaire | through study completion, an average of 1 year
  Potential predictors of the outcome are clinical symptoms. Additional covariables will be patient characteristics including age and gender and disease characteristics. Regression analysis will be used as the main statistical method. Descriptive statistics and graphs and inferential statistics will be used as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- AKH Wien, Vienna, Austria